CLINICAL TRIAL: NCT07047833
Title: Plyometric Training With or Without Hamstring Strengthening for Preventing ACL Injuries in Female Amateur Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Fareeha Raja, Student, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec-UOL-/287/08/24
Record Dates: First submitted 2025-04-04; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: ACL Injuries
Keywords: ACL injury prevention; Plyometric training; Hamstring strengthening; Female athletes; Functional mobility; Dynamic balance
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plyometric Training with Hamstring Strengthening (Experimental): Participants in this group received a six-week intervention consisting of plyometric training combined with targeted hamstring strengthening exercises. Each session was 60 minutes long and conducted twice per week. Plyometric drills included squat jumps, depth jumps, and lateral jumps. Hamstring strengthening included Nordic curls and machine-based leg curls. All participants completed standardized warm-up and cool-down routines. The goal was to assess the additive effect of hamstring strengthening on ACL injury prevention metrics such as strength, balance, and functional mobility.
  Interventions: Behavioral: Plyometric Training with Hamstring Strengthening
- Plyometric Training Only (Experimental): This group received plyometric training only over a six-week period, with sessions lasting 40 minutes and conducted twice weekly. Exercises included squat jumps, depth jumps, and lateral jumps, performed with progressive intensity. Participants underwent a standardized warm-up and cool-down in each session. The purpose of this arm was to evaluate the effectiveness of plyometric training alone in improving strength, balance, and functional mobility for ACL injury prevention.
  Interventions: Behavioral: Plyometric Training Only

INTERVENTIONS:
Behavioral: Plyometric Training with Hamstring Strengthening — This intervention consisted of a six-week training protocol involving both plyometric exercises and targeted hamstring strengthening. Sessions were conducted twice per week, lasting 60 minutes each. Plyometric drills included squat jumps, depth jumps, and lateral jumps, while hamstring exercises included Nordic hamstring curls and machine-based leg curls. All sessions included a standardized 15-minute warm-up and a 5-minute cool-down. The program was designed to enhance lower limb strength, balance, and neuromuscular control for ACL injury prevention in female amateur athletes.
  Arms: Plyometric Training with Hamstring Strengthening
Behavioral: Plyometric Training Only — This intervention involved a six-week plyometric-only training program delivered twice weekly for 40-minute sessions. Exercises included squat jumps, depth jumps, and lateral jumps, performed with progressive intensity and control. Each session included a standardized 15-minute warm-up and a 5-minute cool-down. The program aimed to improve lower limb power, balance, and functional mobility to reduce the risk of ACL injuries in female amateur athletes.
  Arms: Plyometric Training Only

SUMMARY:
This randomized controlled trial explored the effect of plyometric training with or without hamstring strengthening in preventing anterior cruciate ligament (ACL) injuries among female amateur athletes aged 18 to 30. Sixty participants were divided equally into two groups: one received plyometric training combined with hamstring strengthening, and the other received plyometric training only. Both groups trained twice per week over a six-week period. Outcomes measured included knee strength (flexion and extension), dynamic balance (Star Excursion Test), and functional mobility (KOOS).

DETAILED DESCRIPTION:
This study examined whether combining hamstring strengthening with plyometric training provides greater benefits in preventing anterior cruciate ligament (ACL) injuries than plyometric training alone among female amateur athletes. Conducted as a randomized controlled trial, the research involved 60 participants aged 18 to 30, randomly assigned to two equal groups. Group A underwent a six-week intervention involving both plyometric and hamstring strengthening exercises, while Group B participated in plyometric training only. Each group trained twice weekly, and the outcomes were measured at baseline, Week 3, and Week 6 using a handheld dynamometer for knee strength (flexion and extension), the Star Excursion Balance Test (SET) for dynamic balance, and the Knee Injury and Osteoarthritis Outcome Score (KOOS) for functional mobility.

ELIGIBILITY:
Inclusion Criteria:

* Female amateur athletes between the ages of 18-30 years old.
* Participating in sports that involve jumping, cutting and pivoting movements (e.g. basketball, soccer).
* On average, athletes exercised between six and eight times per week including competition.
* Able to perform basic jumping and landing mechanics safely.

Exclusion Criteria:

* Recreational athlete or untrained individual
* Athletes with less than five training sessions per week.
* Athletes who were operated with techniques other than the bone patellar-tendon, bone graft (BPTB), or who were operated by different surgeons and rehabilitated by several physical therapist.
* Athletes with a history of muscle or joint injuries.
* Athletes who had already followed a pre-operative rehabilitation program.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Knee Flexion and Extension Strength (Measured Using Handheld Dynamometer) | Baseline, Week 3, and Week 6
  Lower limb strength was assessed through a handheld dynamometer measuring knee flexion and extension in kilograms. This tool has high reliability for assessing muscle strength and functional performance in athletic populations. Measurements were taken at baseline, Week 3, and Week 6 to evaluate changes over time due to the training interventions.

SECONDARY OUTCOMES:
Dynamic Balance (Assessed Using Star Excursion Balance Test - SEBT) | Baseline, Week 3, and Week 6
  The SEBT evaluates dynamic postural control and balance by measuring reach distance in multiple directions while maintaining single-leg stance. It is a validated predictor of lower extremity injury risk and is used to track neuromuscular improvements in response to training. Performance was recorded at three intervals during the study.
Functional Mobility (Assessed Using KOOS - Knee Injury and Osteoarthritis Outcome Score) | Baseline, Week 3, and Week 6
  The KOOS is a patient-reported outcome tool consisting of 5 subscales: Pain, Symptoms, ADL, Sport/Rec, and Quality of Life. It assesses functional limitations and knee-related quality of life. Scores range from 0 (severe problems) to 100 (no problems). It was used to monitor improvements in knee function due to training.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kasmi S, Zouhal H, Hammami R, Clark CCT, Hackney AC, Hammami A, Chtara M, Chortane SG, Salah FZB, Granacher U, Ounis OB. The Effects of Eccentric and Plyometric Training Programs and Their Combination on Stability and the Functional Performance in the Post-ACL-Surgical Rehabilitation Period of Elite Female Athletes. Front Physiol. 2021 Jul 2;12:688385. doi: 10.3389/fphys.2021.688385. eCollection 2021. PMID 34276409